CLINICAL TRIAL: NCT04256382
Title: Dementia Pain Management Knowledge Scale Development and Impact of an Educational Program on Hospital Nurses' Knowledge Evaluation
Brief Title: Dementia Pain Management Educational Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: KMUHIRB-E(II)-20170072
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The experimental group took two-hour online course about dementia pain care in two weeks.
  Interventions: Other: dementia pain care education
- comparison group (Active Comparator): The comparison group took two-hour online course about dementia care in two weeks.
  Interventions: Other: dementia care education

INTERVENTIONS:
Other: dementia pain care education — Participants are educated about dementia pain care.
  Arms: experimental group
Other: dementia care education — Participants are educated about dementia pain care.
  Arms: comparison group

SUMMARY:
This study aims to develop and test a scale for exploring hospital nurses' knowledge about dementia pain and dementia pain management.

DETAILED DESCRIPTION:
The researcher recruited 285 nurses from three hospitals, and divided them into the experimental group and the comparison group. The experimental group took two-hour online course about dementia pain care in two weeks. The comparison group took two-hour online course about dementia care in two weeks. The nurses performed a post-test after the two-week course immediately; two weeks later, the second post-test was performed again.

ELIGIBILITY:
Inclusion Criteria:

* Nurses working in district hospitals, regional hospitals, or medical centers.

Exclusion Criteria:

* Nurses working with obstetrics, pediatrics, or outpatient.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2019-12-24 (Actual); Study Completion 2020-02-03 (Actual)

PRIMARY OUTCOMES:
score of Dementia Pain Management Knowledge Scale | 2 months
  Testing nurses' Dementia Pain Management Knowledge. The minimum value of this scale is 15, and the maximum value is 0. Higher scores mean having better Dementia Pain Management Knowledge.

SECONDARY OUTCOMES:
score of Dementia Care Knowledge 16 | 2 months
  Testing nurses' Dementia Care Knowledge. The minimum value of thus scale is 16, and the maximum value is 0. Higher scores mean having better Dementia Care Knowledge.
score of the Chinese version of the Knowledge and Beliefs About Pain in Elderly Patients With Dementia (KBPED-C) questionnaire | 2 months
  Testing nurses' Knowledge and Beliefs About Pain in Elderly Patients With Dementia. The minimum value of this scale is 85, and the maximum value is 17. Higher scores mean having better Knowledge and Beliefs About Pain in Elderly Patients With Dementia.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan